CLINICAL TRIAL: NCT07342842
Title: Comparison of the Ultrasonic Cardiac Output Monitor and Echocardiography for Hemodynamic Assessment in Pediatric Anesthesia: A Prospective Observational Study
Brief Title: Comparison of the Ultrasonic Cardiac Output Monitor and Echocardiography for Hemodynamic Assessment in Pediatric Anesthesia
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Volkan Kuzlu, principal investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: USCOM-Echo
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2021-03

CONDITIONS: USCOM; Echocardiography; Echocardiography Guided Fluid Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: USCOM — Ultrasound cardiac output monitoring is performed using a suprasternal approach to obtain spectral Doppler signals from the ascending aorta. After anesthesia induction and stabilization, the probe is positioned at the suprasternal notch to acquire optimal Doppler waveforms. Velocity time integral (VTI), stroke volume (SV), cardiac output (CO), stroke volume variation (SVV), systemic vascular resistance (SVR), and device-calculated aortic valve area (AVA) are recorded using the manufacturer's algorithm. Only high-quality Doppler envelopes are accepted, and measurements are repeated if artifacts or poor signal quality are present. All parameters are obtained consecutively under unchanged ventilatory and hemodynamic conditions.
Other: Echocardiography — Transthoracic echocardiography is performed immediately after USCOM measurements under unchanged anesthetic depth, ventilator settings, and patient positioning. Using a pediatric probe, suprasternal Doppler recordings are obtained from the ascending aorta, with the Doppler cursor aligned as parallel as possible to blood flow; angle correction is applied when necessary. Velocity time integral (VTI) is measured from the largest and most clearly defined spectral Doppler envelope. The aortic annulus diameter is obtained from the parasternal long-axis view during midsystole, and aortic valve area is calculated. Stroke volume is derived as aortic valve area × VTI, and cardiac output is calculated as stroke volume × heart rate. Inspiratory and expiratory VTI values are recorded to determine respiratory variation and calculate stroke volume variation. Each parameter is measured three times and averaged for analysis.

SUMMARY:
This prospective observational pilot study evaluates agreement between Ultrasound Cardiac Output Monitor (USCOM) measurements and transthoracic echocardiography-derived hemodynamic parameters in pediatric patients under standardized general anesthesia prior to surgical incision. Under stable hemodynamic and ventilatory conditions, suprasternal Doppler-derived velocity time integral (VTI), stroke volume (SV), cardiac output (CO), stroke volume variation (SVV), and aortic valve area (AVA) are obtained sequentially with USCOM and echocardiography within a short time window without changes in ventilation, anesthetic depth, positioning, fluid therapy, or vasoactive support. Agreement is assessed using correlation and Bland-Altman analyses.

DETAILED DESCRIPTION:
This prospective observational pilot study is designed to evaluate the agreement between Ultrasound Cardiac Output Monitor (USCOM) measurements and transthoracic echocardiography-derived hemodynamic parameters in pediatric patients undergoing elective surgery under standardized general anesthesia.

After anesthesia induction and airway management, patients are allowed to reach stable hemodynamic and ventilatory conditions. Heart rate, noninvasive blood pressure, peripheral oxygen saturation, tidal volume, respiratory rate, and positive end-expiratory pressure are documented to confirm comparable physiological conditions during all measurements.

All measurements are performed before surgical incision and under unchanged ventilator settings, anesthetic depth, and patient positioning. No fluid administration, vasoactive medication, or ventilatory adjustments are made between techniques.

USCOM measurements are obtained first using a suprasternal approach to acquire spectral Doppler signals. Device-derived parameters, including velocity time integral (VTI), stroke volume (SV), cardiac output (CO), stroke volume variation (SVV), systemic vascular resistance (SVR), and device-calculated aortic valve area (AVA), are recorded consecutively during spontaneous or controlled mechanical ventilation without apnea. Only Doppler signals with clearly defined spectral envelopes are accepted. Measurements with artifacts or poor signal quality are repeated until optimal tracings are achieved.

Immediately afterward, transthoracic echocardiography is performed using a pediatric probe. Suprasternal Doppler recordings are aligned as parallel as possible to blood flow in the ascending aorta, and angle correction is applied when required. VTI is measured from the largest and most clearly defined spectral Doppler envelope. The aortic annulus diameter is obtained from the parasternal long-axis view during midsystole, and aortic valve area is calculated. Stroke volume is derived as aortic valve area × VTI, and cardiac output is calculated as stroke volume × heart rate. Inspiratory and expiratory VTI values are recorded to determine respiratory variation and calculate SVV.

USCOM and echocardiography measurements are performed sequentially within a 1-2-minute time window to minimize the impact of temporal hemodynamic variability. Each parameter is measured three consecutive times, and the average value is used for statistical analysis.

All examinations are conducted by a single experienced operator who completed supervised echocardiography training and independently performed at least 30 validated measurements before study initiation to minimize interobserver variability.

The primary objective is to assess agreement between USCOM and echocardiography for stroke volume and cardiac output measurements. Secondary objectives include correlation of suprasternal VTI values, agreement in SVV measurements, comparison of USCOM-calculated versus echocardiography-derived aortic valve area, and Bland-Altman analysis of all paired hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6 months to 15 years
* ASA physical status I-II
* Scheduled for elective surgery requiring general anesthesia
* Written informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

* Intracardiac or extracardiac shunts
* Aortic valve disease
* Anatomical limitation preventing suprasternal Doppler assessment
* Required Doppler angle correction >20° during echocardiography evaluation
* Emergency surgery
* Inability to obtain informed consent

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 6 months to 15 years with ASA physical status I-II who are scheduled for elective surgery requiring general anesthesia. All participants undergo noninvasive suprasternal Doppler and transthoracic echocardiography measurements under standardized anesthetic conditions before surgical incision.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Agreement Between USCOM and Echocardiography for Stroke Volume and Cardiac Output | Intraoperative, after induction and stabilization and before surgical incision (single assessment; within 1-2 minutes between methods).
  Agreement of paired SV and CO values obtained by USCOM and echocardiography under stable conditions, evaluated using Bland-Altman analysis (bias and 95% limits of agreement) and correlation.

SECONDARY OUTCOMES:
Correlation Between USCOM VTI and Echocardiography VTI (Suprasternal Doppler) | Single intraoperative assessment after induction and stabilization and before surgical incision (measurements obtained sequentially within 1-2 minutes).
  To evaluate the strength of association between velocity time integral (VTI) values obtained using suprasternal Doppler with USCOM and those measured by transthoracic echocardiography under stable anesthetic and ventilatory conditions.
Agreement Between USCOM and Echocardiography for Stroke Volume Variation | Single intraoperative assessment after induction and stabilization and before surgical incision (measurements obtained sequentially within 1-2 minutes).
  To assess agreement between USCOM-derived and echocardiography-derived stroke volume variation (SVV) values calculated from inspiratory and expiratory Doppler measurements using paired Bland-Altman analysis and correlation methods.
Comparison of Device-Calculated Versus Echocardiography-Derived Aortic Valve Area | Single intraoperative assessment after induction and stabilization and before surgical incision (measurements obtained sequentially within 1-2 minutes).
  To compare aortic valve area (AVA) values automatically calculated by USCOM using biometric algorithms with AVA values derived from echocardiographic aortic annulus measurement and Doppler velocity time integral.
Bland-Altman Agreement of Paired Hemodynamic Variables | Single intraoperative assessment after induction and stabilization and before surgical incision (measurements obtained sequentially within 1-2 minutes).
  To evaluate agreement between USCOM and echocardiography for paired hemodynamic variables, including stroke volume, cardiac output, velocity time integral, stroke volume variation, and aortic valve area, using Bland-Altman analysis with calculation of bias and limits of agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided